CLINICAL TRIAL: NCT02836860
Title: Effects of Adding Tactile Stimuli to Verbal Instructions for Lumbar Multifidus Muscle Activation in Healthy Adults and Patients With Low Back Pain
Brief Title: Effects of Tactile Stimuli for Lumbar Multifidus Muscle Activation in Healthy Adults and Patients With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Sharon Wang-Price, Professor, Texas Woman's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17920
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Controls (Other): Effects of tactile stimulation on lumbar multifidus activation in healthy adults without LBP.
  Interventions: Other: Tactile stimuli
- Low Back Pain (Other): Effects of tactile stimulation on lumbar multifidus activation in adults with LBP.
  Interventions: Other: Tactile stimuli

INTERVENTIONS:
Other: Tactile stimuli — Both groups will receive tactile stimuli: hand touch on the right and left lumbar multifidus muscles at L4-5

SUMMARY:
The purpose of this study is to compare combined tactile stimulation and verbal instruction to verbal instruction only on lumbar multifidus muscle activation in asymptomatic healthy adults and in patients with LBP.

DETAILED DESCRIPTION:
Reduced lumbar multifidus muscle contraction has been observed in patients with low back pain (LBP). Currently, considerable evidence supports spinal stabilization exercises for treating LBP, including lumbar multifidus muscle activation exercises. Clinicians often apply a tactile stimulation on the muscle in addition to verbal instructions to ensure muscle activation. However, whether or not the addition of tactile stimulation would increase muscle activation has not been studied. Therefore, the investigators plan to use electromyography (EMG) to examine if addition of tactile stimulation to verbal instructions would increase lumbar multifidus muscle activation in healthy adults and patients with LBP.

The purpose of this study is to compare combined tactile stimulation and verbal instruction to verbal instruction only on lumbar multifidus muscle activation in asymptomatic healthy adults and in patients with LBP. The research hypothesis is that the lumbar multifidus muscle activation will be increased when the participants are given combined tactile stimulation and verbal instruction as compared to when the participants are given verbal instruction only.

Participants:

Eligible participants are English-speaking adults 18 years of age or older. Additional criteria for asymptomatic healthy adults include no existing LBP and no LBP in the past year. Additional criteria for patient participants include existing LBP near the L5-S1 level with an average pain intensity score ≥ 2/10 in the past 24 hours (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain). Exclusion criteria for all participants include previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis), cancer of the lower quadrant, neurological disorders, allergic reaction to ultrasound gel, or inability to obtain testing positions (prone lying).

The investigators plan to enroll 20 asymptomatic healthy adults, and 20 patients with LBP. Potential participants will be recruited from the local community (including but not limited to Texas Woman's University - Dallas) via flyers. The flyers will be posted at the TWU - Dallas campus and other community centers with approval. Participants who are interested in taking part in the study will be asked to call investigators to schedule an appointment time for testing. The consent form will be presented at the beginning of the appointment.

Procedures:

After participants are informed of the risks, benefits and procedures of the study, they will be asked to sign a written consent form approved by the TWU Institutional Review Board - Dallas. Eligible participants will be asked to complete an intake form, asking them about their age, gender, and past medical history. For participants with existing low back pain, they will be asked about their pain location, duration, intensity, and nature, medicine use of their existing LBP and their LBP history.

Instrumentation

1. The Modified Oswestry Low Back Pain Index (OSW) questionnaire will be used to determine an individual's perceived disability and function limitation due to his/her low back pain. The OSW questionnaire has been shown to be reliable and valid.
2. A Delsys EMG system with 2 wireless surface electrodes (Delsys Inc., Boston, MA) will be used to obtain muscle activities. The bandwidth of the EMG system will be set at 20 to 450 Hz with a gain of 1,000. The EMG signal will be recorded at a sampling rate of 1,000 Hz. Each surface electrode has a built-in reference electrode.

EMG Recording Prior to EMG recording, the anatomy and location of the lumbar multifidus muscle will be explained and shown to participants using a model and pictures. Next, participants will lie in prone on an examination table with their arms on the sides. A pillow will be placed under the participant's abdomen to flatten the lumbar lordotic curve and an inclinometer will be placed on the lumbosacral junction to ensure the lumbar curve ≤10 degrees. The spinous processes of the L4-S2 and sacral sulcus will be identified by palpation and marked with an erasable pen.

Next, one investigator will prepare the participant's skin in the areas of the 2 electrode placements. The skin will be cleaned with isopropyl alcohol. If there is excessive hair, a new disposable razor will be used to shave the hair to improve the quality of the EMG recording. If shaving is required, the investigator will wear gloves to perform shaving following universal precautions. Once the skin is prepared for EMG recording, 2 electrodes will be placed on the skin over the right and left lumbar multifidus at two at the L4-5 level.

The EMG of lumbar multifidus will be recorded 3 times "at rest" first prior to each of muscle activation conditions: (1) verbal instruction only, and (2) combined tactile stimulation and verbal instruction. For both the muscle activation conditions, the participant will be asked to assume a starting position: abduct the contralateral shoulder and flex the contralateral elbow to approximately 90°. The contralateral side will be opposite to the painful side of patients with LBP or the left side of the asymptomatic participants. If the patient has bilateral LBP, the contralateral side will be the less painful side.

During verbal instruction, one investigator will give a verbal instruction and then ask the participant to perform a contralateral-arm task, in which the participant will lift the contralateral arm approximately 5 cm above the table and hold for 5 seconds. The verbal instruction was selected based on our published pilot study which showed that this instruction seemed to activate lumbar multifidus muscle the most: "Breathe normally, without moving the pelvis or spine, think about tilting the pelvis forward without actually moving it, and lift the left (right) arm".

During tactile stimulation, the investigator will place his/her middle 2 or 3 fingers on the lumbar multifidus at L5-S1 between the 2 electrodes before the verbal instruction is given. The investigator will then give the same verbal instruction and ask the participant to perform the contralateral-arm-lift task while maintaining finger contact on the multifidus muscle during muscle activation. EMG testing will start after the verbal instruction is completed.

For each muscle activation condition, participants will hold each contraction for 5-8 seconds, and a 10-minute rest will be given between the 2 contraction conditions.

ELIGIBILITY:
Inclusion Criteria:

* Additional criteria for asymptomatic healthy adults include no existing LBP and no LBP in the past year. Additional criteria for patient participants include existing LBP near the L5-S1 level with an average pain intensity score ≥ 2/10 in the past 24 hours (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain).

Exclusion Criteria:

* Exclusion criteria for all participants include previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis), cancer of the lower quadrant, neurological disorders, allergic reaction to ultrasound gel, or inability to obtain testing positions (prone lying).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Electromyographic (EMG) amplitude | 8 seconds, 5 repetitions during one visit
  Surface EMG activity of the right and left lumbar multifidus at L4-5 level

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No